CLINICAL TRIAL: NCT00053261
Title: Vaginal Length, Elasticity, Lubrication And Sexual Function In Women With Stage IB2 Cervix Carcinoma
Brief Title: Vaginal Changes and Sexual Function in Patients With Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Other Study IDs: CDR0000269327; GOG-8003
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2005-06

CONDITIONS: Cervical Cancer; Sexuality and Reproductive Issues
Keywords: sexuality and reproductive issues; stage IB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sexuality

INTERVENTIONS:
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Vaginal changes that may effect sexual function occur in patients undergoing treatment for cervical cancer.

PURPOSE: Clinical trial to determine the type of vaginal changes such as vaginal dryness that occur in patients receiving treatment for cervical cancer and the effect these changes have on sexual function.

DETAILED DESCRIPTION:
OBJECTIVES:

* Obtain estimates of changes in vaginal length, perceived vaginal elasticity, perceived vaginal lubrication, and sexual activity, response, and satisfaction among patients with stage IB2 cervical cancer.
* Compare these differences between the patients in the two treatment groups in GOG-0201.
* Determine the relationships between vaginal dilation activities and vaginal length changes in these patients.
* Determine the association between smoking and vaginal length and between smoking and vaginal dryness in these patients after therapy for cervical cancer.
* Assess the extent of subject interest in and preferred methods of sexual counseling related to problems resulting from treatment in these patients.

OUTLINE: Vaginal length is measured using Vaginal Sound, a modified plastic vaginal dilator. The data about vaginal elasticity and lubrication and sexual activity, response, and satisfaction are obtained from patient self-report, as well as vaginal dilation activities. Measurement and assessments are taken before treatment and then at 3, 6, 12, and 24 months.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: Approximately 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Entered and treated on GOG-0201 or eligible for and treated on either arm of GOG-0201

  * May have refused entry on GOG-0201 as long as treatment is prescribed according to one or the other arm

PATIENT CHARACTERISTICS:

Age

* Under 70

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Watkins Bruner, RN, PhD, Study Chair — Fox Chase Cancer Center
Locations (12):
- United States (12):
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania